CLINICAL TRIAL: NCT06140199
Title: Comparing Minimally Invasive Treatments for Pilonidal Disease: LA POPA Trial (Laser And Pit-picking OR Pit-picking Alone)
Acronym: LA POPA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: dr. IJM Han-Geurts (Other)
Collaborators: Flevoziekenhuis (Other); Proctos Kliniek (Other); Sint Jans Gasthuis Weert (Unknown); UMC Utrecht (Other); Ziekenhuis Amstelland (Other); Treant ziekenhuis (Unknown); Albert Schweitzer Hospital (Other)
Responsible Party: Sponsor-Investigator, dr. IJM Han-Geurts, Local investigator, Proctos Kliniek
Organization: Proctos Kliniek (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL84679.018.23
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Pilonidal Sinus; Pilonidal Disease; Pilonidal Sinus of Natal Cleft; Pilonidal Disease of Natal Cleft; Pilonidal Sinus Without Abscess
Keywords: Pit-picking; Laser-assisted therapy; SiLaC; Minimally invasive surgery
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Intervention Model Description: Multicentre, single-blinded, randomised, controlled, superiority trial. It
Who Masked: Outcomes Assessor
Masking Description: Only the outcome assessor is blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pit-picking surgery (Active Comparator)
  Interventions: Procedure: Pit-picking surgery
- Pit-picking surgery with Sinus Laser assisted Closure (Experimental)
  Interventions: Procedure: Pit-picking surgery with Sinus Laser assisted Closure

INTERVENTIONS:
Procedure: Pit-picking surgery — Patients are placed in left-side position. After shaving, cleaning and scrubbing of the skin with alcoholic chlorhexidine, double strong tape is placed on the right buttock in order to increase exposure. Local anaesthesia is administered before incision with 20 ml xylocaine or lidocaine 1-2%. In principle, all sinusoidal pits are cut out with a margin of at least 1 mm with a biopsy core punch (4 mm, 6 mm or 8 mm depending on pit size) or an oval excision of the pits is performed. Hair and debris is removed from the sinus tracts with a small surgical spoon or mosquito clamp. Rigorous de-epithelialisation of the underlying sinus is performed with the spoon through every pit, whilst removing even more debris and hairs. At the end of the procedure a debris washout is performed with saline solution, the wounds are left open for secondary healing and sterile dressings are applied.
  Arms: Pit-picking surgery
Procedure: Pit-picking surgery with Sinus Laser assisted Closure — The pit picking procedure is described above. Subsequently, a radial diode laser probe at 1470 nm wavelength is used for delivering homogeneous (360 degrees) energy to the surrounding epithelium. The laser energy is 13 Joule, given continuously. First, a 'preparatory laser treatment' is performed to extract any missed hairs or debris, after which the sinus tracts are cleansed with a surgical spoon again. During the following definitive procedure, the probe is withdrawn at an approximate speed of 1 cm per three seconds, causing the small sinus tracts to shrink and close. Large sinus tracts remain open because very large sinus tracts or cavities cannot be closed with the 3mm laser fibre. The injury to the endothelium will cause granulation and create oedema for collapsing of the tract. The remaining open wounds are left open for secondary healing and sterile dressings are applied.
  Arms: Pit-picking surgery with Sinus Laser assisted Closure

SUMMARY:
The goal of this randomized clinical trial is to establish the efficacy of 'pit picking with laser therapy' versus 'pit picking alone' on both short and long-term outcomes in patients of 12 years and older with primary pilonidal sinus disease.

The main questions it aims to answer are:

* The overall success rate of treatment which is defined as: closure of all pits at 12 months of follow-up.
* Secondary endpoints: succes rat eof treatment during long-term follow-up, wound closure time, pain scores, complication rate, work rehabilitation, time to return to daily activities, quality of life, persisting complaints, patient satisfaction, costs and the need for secondary or revision surgery.

Participants will allocated to pit picking alone or combined with lasertherapy.

The extra burden for participating patients is expected to be minimal to moderate. Participants will have two extra hospital visits in casethey are enrolled in our study: 6 and 12 months after enrolment. Postoperatively the normal scheme of follow up appointments wil be used: 2 and 6 weeks after treatment at the outpatient clinic of the treating surgeon. A telephone appointment with the researcher will be scheduled 4 weeks after treatment. Patients are asked to complete questionnaires at various time points, which will be sentto them by email and will take approximately 5-10 minutes each time. The content includes general and disease specific Quality of Life (QoL) questionnaires. The investigators do not expect any extra adverse reactions or events in respect to participation in the study because both procedures are considered standard of care in the participating clinics. However, because both interventions are surgical procedures a small percentage of adverse events or postoperative complications can be expected.

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 12 years and older who present with primary pilonidal sinus disease; Type 1b and 3 of the Dutch staging system
* Obtained written informed consent by the patient and/or legal representative/parent
* Sufficient understanding of the Dutch written language (reading and writing)
* Eligible for questionnaires sent by e-mail

Exclusion Criteria:

* Asymptomatic (Type 1a), recurrent (Type 4; except those patients who only have had drainage of their abscess and no other surgical treatment), or chronic wounds (hypergranulating) after PSD surgery (Type 5) of the Dutch staging system
* Patients with known underlying or concomitant medical conditions that may interfere with normal wound healing (e.g. systemic skin and connective tissue diseases, any kind of congenital defect of metabolism including insulin-dependent diabetes mellitus, Cushing syndrome or disease, scurvy, chronic hypothyroidism, congenital or acquired immunosuppressive condition, chronic renal failure, or chronic hepatic dysfunction (Child-Pugh class B or C), severe malnutrition, or other concomitant illness which, in the opinion of the investigator, has the potential to significantly delay wound healing)
* Severe drug abuse (and therefore protocol deviation can be expected)
* Patients expected not to comply with the study protocol (including patients with severe cognitive dysfunction/impairment and severe psychiatric disorders)
* Patients with insufficient knowledge of the Dutch written language who are thus unable to answer the questionnaires
* Patients that are unable or not willing to give full informed consent

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 482 (Estimated)
Dates: Start 2024-08-28 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2032-05 (Estimated)

PRIMARY OUTCOMES:
Succes rate of treatment | 1 year
  Success rate of treatment, defined as closure of all pits at 1 year follow-up. Closure of the pits will be assessed by the treating surgeon by means of an extensive physical examination.

SECONDARY OUTCOMES:
Success rate of treatment at long-term follow-up | 3-5 years
  Success rate of treatment at 3 and 5 years follow up
Pain score | 6 weeks
  Pain scores in the period after surgery (VAS). VAS score scale: 0-10, higher score meaning a worse outcome.
Patient reported outcome measures | 5 years
  PROMs, defined as persisting complaints: itching, wound fluid leakage, blood loss, pus, pain, social burden (shame/embarrassment). PROMs will be scored on a scale: 1-5, with a higher score meaning a worse outcome.
Wound healing and complications | 1 year
  Wound and complications
Work rehabilation | 6 weeks
  Work rehabilitation; number of days
Return to daily activities | 6 weeks
  Time until return to daily activities; number of days
Recurrence rate | 5 years
  Recurrence rate at 1, 3 and 5 years of follow-up
Need for secondary or revision surgery | 5 years
  Need for seondary or revision surgery for pilonidal disease
Patient satisfaction | 5 years
  Patient satisfaction with treatment (scored on a likert scale 0-10, with a higher score meaning a better outcome)
Quality adjusted life years (QALYs) | 5 years
  Quality of life after treatment (Eq-5d-5l; will be converted to Quality adjusted life years (QALYs; range 0-1, with 1 the highest score and the better outcome)
Absence of symptoms | 1 year
  Absence of symptoms at 1-yars follow-up: participants will be asked a dichotomous question during their 1-year follow-up appointment. At that moment, do they feel their symptoms from pilonidal sinus disease are: A) cured or improved when compared with before treatment? or B) unchanged or worse when compared with before treatment?

CONTACTS AND LOCATIONS:
Overall Officials: Robert Smeenk, MD PhD, Principal Investigator — Albert Schweitzer Hospital

IPD SHARING:
Plan to Share IPD: No
On reasonable request.

REFERENCES:
- [Result] Sluckin TC, Hazen SJA, Smeenk RM, Schouten R. Sinus laser-assisted closure (SiLaC(R)) for pilonidal disease: results of a multicentre cohort study. Tech Coloproctol. 2022 Feb;26(2):135-141. doi: 10.1007/s10151-021-02550-4. Epub 2022 Jan 7. PMID 34993686